CLINICAL TRIAL: NCT01091714
Title: Is Omega-3 Fatty Acid RBC Saturation Product Dependent?
Brief Title: Is Omega-3 Fatty Acid Red Blood Cell (RBC) Saturation Product Dependent?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bucci Laser Vision Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01-2010; NCT01173185 (obsolete NCT alias)
Record Dates: First submitted 2010-03-18; First posted 2010-03-24 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Cardioprotective Levels
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PRN Dry Eye Omega Benefits (Active Comparator): 4 capsules per day = 2240 mg Omega-3s
  Interventions: Dietary Supplement: Omega-3
- Nature's Made (Active Comparator): 2 capsules per day = 2400mg Omega-3s
  Interventions: Dietary Supplement: Omega-3
- Thera Tears (Active Comparator): 4 capsules per day = 2332mg Omega-3s
  Interventions: Dietary Supplement: Omega-3

INTERVENTIONS:
Dietary Supplement: Omega-3 — Approximately 2400 mg of Omega-3s taken once daily by capsule, taken for the duration of the study.
  Arms: Nature's Made
Dietary Supplement: Omega-3 — Approximately 2240 mg of Omega-3s taken once daily by capsule, taken for the duration of the study.
  Arms: PRN Dry Eye Omega Benefits
Dietary Supplement: Omega-3 — Approximately 2332 mg of Omega-3s taken once daily by capsule, taken for the duration of the study.
  Arms: Thera Tears

SUMMARY:
To demonstrate that RBC saturation of the Omega-3 fatty acids reaching cardioprotective levels as proven with the HS-Omega-3 Index test will be achieved most efficiently depending on a specific product utilized within this study.

DETAILED DESCRIPTION:
To demonstrate that RBC saturation of the Omega-3 fatty acids reaching cardioprotective levels as proven with the HS-Omega-3 Index test will be achieved most efficiently depending on a specific product utilized within this study. The HS-Omega-3 Index is a new test that measures blood levels of the cardioprotective omega-3 fatty acids, EPA and DHA. RBS saturation is being measured to identify how much Omega 3 is in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent.
* Subject motivation and willingness to cooperate with the investigator by following the required medication regimen.
* Subject willingness and ability to return for all visits during the study.
* Must be willing to discontinue all use of Omega-3 supplementation 2 weeks prior to study participation.

Exclusion Criteria:

* Concurrent involvement in any other clinical trial involving an investigational drug or device.
* Compromised cognitive ability which may be expected to interfere with study compliance.
* Uncontrolled or poorly controlled systemic disease ot the presence of any significant illness that could, in the judgment of the investigator, jeopardize subject safety or interfere with the interpretation of the results of the study.
* Subjects must not eat more that 1 non-fried fish meal per week.
* Subjects must not have undergone any bariatric surgery or have a malabsorption disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
RBC saturation of Omega-3 fatty acids reaching cardioprotective levels as proven with HS-Omega_3 Index test. | one month

SECONDARY OUTCOMES:
RBC saturation of Omega-3 fatty acids reaching cardioprotective levels as proven with HS-Omega_3 Index test. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Bucci, Jr., MD, Principal Investigator — Bucci Laser Vision Institute
Locations (1):
- Bucci Laser Vision Institute, Wilkes-Barre, Pennsylvania, United States